CLINICAL TRIAL: NCT05323240
Title: Repeated Exposure Study
Brief Title: Health Effects of Repeated Exposure to Low Levels of Concentrated Ambient Particles in Healthy Young Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: U.S. EPA Human Studies Facility (U.S. Federal Agency)
Responsible Party: Principal Investigator, Haiyan Tong, Principal Investigator, U.S. EPA Human Studies Facility
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RPTCAP
Record Dates: First submitted 2021-11-29; First posted 2022-04-12 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Air Pollution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filtered air exposure (Experimental): Subjects will be randomly exposed to three consecutive days of filtered air exposure arm in a double-blind cross-over fashion in an exposure chamber, and exposures will be separated by a minimum of 13 days from the PM2.5 arm.
  Interventions: Other: Filtered air exposure
- PM exposure (Experimental): Subjects will be randomly exposed to three consecutive days of PM2.5 exposure arm in a double-blind cross-over fashion in an exposure chamber, and exposures will be separated by a minimum of 13 days from the filtered air arm.
  Interventions: Other: PM exposure

INTERVENTIONS:
Other: PM exposure — To determine whether 3-day consecutive exposures to levels of fine particulate matter (PM2.5) that are close to the current 24-hr national standard will cause changes in inflammatory and cardiopulmonary endpoints.
  Arms: PM exposure
Other: Filtered air exposure — To determine whether 3-day consecutive exposures to filtered air will cause changes in inflammatory and cardiopulmonary endpoints.
  Arms: Filtered air exposure

SUMMARY:
Purpose: To determine whether 3-day consecutive exposures to levels of fine particulate matter (PM2.5) that are close to the current 24-hr national standard will cause changes in inflammatory and cardiopulmonary endpoints in healthy young individuals.

Participants: 20 healthy males and females aged 18-35 years.

Procedures (methods): Subjects will be randomly exposed to three consecutive days of filtered air (4 hr/day) and three consecutive days of PM2.5 (approximately 35 µg/m3; 4 hr/day) in an exposure chamber. Blood collection for inflammatory factors such as C-reactive protein (CRP), clotting factors; heart rate variability (HRV); spirometry; and a symptom questionnaire will be conducted before and after each exposure.

ELIGIBILITY:
Inclusion Criteria:

1. . Age 18-35 years old healthy male and female (BMI values between 19 and 30).
2. . Physical conditioning allowing intermittent, moderate exercise for 2 hours, and ability to complete the exposure exercise regimen to induce a minute ventilation rate of 20 L/min/m2 for 15 min without exceeding 80% of projected maximal heart rate. Predicted maximal heart rate will be calculated using the equation [described by Tanaka et al.: (2001) J. Am. Coll. Cardiol: 208bpm-((0.7) x (age in years))]
3. . Normal baseline 12-lead EKG.
4. . Normal lung function based on NHANES III reference values. i. Forced vital capacity (FVC) ≥ 80% of that predicted for age, gender, ethnicity, and height.

   ii. Forced expiratory volume in one second (FEV1) ≥ 80% of that predicted for age, gender, ethnicity, and height.

   iii: FEV1/FVC ratio ≥ 80% of predicted values.
5. . Oxygen saturation greater than 94% at the time of physical exam.

Exclusion Criteria:

1. . Individuals with a diagnosis of COVID-19 and/or hospitalized for COVID-19.
2. . Individuals not vaccinated for COVID-19, or, not 14 days beyond the final dose of receiving a COVID-19 vaccine.
3. . Individuals with a history of acute or chronic cardiovascular disease, chronic respiratory disease, diabetes, rheumatologic diseases, or immunodeficiency state.
4. . Individuals with a CVD risk score greater than 10% using the ACC/AHA ASCVD risk calculator (based on the 10-year risk of heart disease or stroke using the Atherosclerotic Cardiovascular Disease algorithm published in 2013 American College of Cardiology/American Heart Association Guideline on the Assessment of Cardiovascular risk.
5. . Individuals with asthma and a history of asthma.
6. . Individuals who are allergic to chemical vapors or gases.
7. . Females who are pregnant, attempting to become pregnant, or breastfeeding.
8. . Individuals who are currently smoking (including vaping, hookah, e-cigarette) or have a smoking history within 1 year of study.
9. . Individuals living with a smoker who smokes inside the house.
10. . Individuals with a body mass index (BMI) >30 or <19. Body mass index is calculated by dividing the weight in kilograms by the square of the height in meters.
11. . Individuals with occupational exposures to high levels of vapors, dust, gases, or fumes on an on-going basis.
12. . Individuals with uncontrolled hypertension (>140 systolic or >90 diastolic).
13. . Individuals who do not understand or speak English.
14. . Individuals who are unable to perform the exercise required for the study.
15. . Individuals with a history of skin allergies to adhesives used in securing EKG electrodes.
16. . Individuals with unspecified diseases, conditions, or medications that might influence the responses to the exposures, as judged by the medical staff.
17. . Individuals who are unwilling or unable to stop taking over-the-counter pain medications such as aspirin, ibuprofen (Advil, Motrin), naproxen (Aleve), or other non-steroidal anti-inflammatory ("NSAID") medications for 48 hours prior to the exposures and post-exposure visits. Individuals taking vitamins or supplements that the investigators believe may impact the results of the study who are unwilling or unable to stop taking them for at least two weeks before the study. Those not specifically mentioned here may be reviewed by the investigators prior to an individual's inclusion in the study.
18. . Individuals taking systemic steroids or beta-blocker medications.
19. . Individuals with a hemoglobin A1c (HbA1c) level > 6.4%.
20. . Individuals who are claustrophobic.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Blood inflammation marker, CRP, will be measured 2 hours before each air exposure day and follow up day in 20 subjects | Four days
  Venous blood will be collected for CRP measurement 2 hours before each air exposure day on day 1, day 2, day 3, and follow up day in 20 subjects.
Blood inflammation marker, CRP, will be measured 2 hours before each PM exposure day and follow up day in 20 subjects | Four days
  Venous blood will be collected for CRP measurement 2 hours before each PM exposure day on day 1, day 2, day 3 and follow up day in 20 subjects.
Blood inflammation marker, CRP, will be measured 1 hour after each air exposure day in 20 subjects | Three days
  Venous blood will be collected for CRP measurement 1 hour after each air exposure day on day 1, day 2, and day 3 in 20 subjects.
Blood inflammation marker, CRP, will be measured 1 hour after each PM exposure day in 20 subjects | Three days
  Venous blood will be collected for CRP measurement 1 hour after each PM exposure day on day 1, day 2, and day 3 in 20 subjects.

SECONDARY OUTCOMES:
Spirometry will be measured 1 hour before each air exposure day and follow up day in 20 subjects | Four days
  FEV1 and FVC will be measured by spirometry 1 hour before each air exposure day on day 1, day 2, day 3, and follow up day in 20 subjects.
Spirometry will be measured 1 hour before each PM exposure day and follow up day in 20 subjects | Four days
  FEV1 and FVC will be measured by spirometry 1 hour before each PM exposure day on day 1, day 2, day 3 and follow up day in 20 subjects.
Ambulatory ECG will be measured 2 hours before each air exposure day and follow up day in 20 subjects | Four days
  ECG QT interval and frequency power of ECG will be measured by Holter monitor for 5 minutes at 2 hour before each air exposure day on day 1, day 2, day 3, and follow up day in 20 subjects.
Ambulatory ECG will be measured 2 hours before each PM exposure day and follow up day in 20 subjects | Four days
  ECG QT interval and frequency power of ECG will be measured by Holter monitor for 5 minutes at 2 hours before each PM exposure day on day 1, day 2, day 3, and follow up day in 20 subjects.
Spirometry will be measured 1 hour after each air exposure day in 20 subjects | Three days
  FEV1 and FVC will be measured by spirometry 1 hour after each air exposure day on day 1, day 2, and day 3 in 20 subjects.
Spirometry will be measured 1 hour after each PM exposure day in 20 subjects | Three days
  FEV1 and FVC will be measured by spirometry 1 hour after each PM exposure day on day 1, day 2, and day 3 in 20 subjects.
Ambulatory ECG will be measured 2 hours after each air exposure day in 20 subjects | Three days
  ECG QT interval and frequency power of ECG will be measured by Holter monitor for 5 minutes at 2 hours after each air exposure day on day 1, day 2, and day 3 in 20 subjects.
Ambulatory ECG will be measured 2 hours after each PM exposure day in 20 subjects | Three days
  ECG QT interval and frequency power of ECG will be measured by Holter monitor for 5 minutes at 2 hours after each PM exposure day on day 1, day 2, and day 3 in 20 subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States